CLINICAL TRIAL: NCT07122778
Title: Impact of Diet-induced Change in Energy Balance on Metabolism in Endurance Athletes: the Carpe DIEM Study
Brief Title: Impact of Diet-induced Change in Energy Balance on Metabolism in Endurance Athletes
Acronym: Carpe DIEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Royal Centre for Defence Medicine (Other Government)
Responsible Party: Principal Investigator, Josh Bakker-Dyos, Principal Investigator, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 6854-11590; 345572 (Other: Health Research Authority)
Record Dates: First submitted 2025-04-14; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Energy Balance; Energy Deficit; Low Energy Availability; Relative Energy Deficiency in Sport
Keywords: energy deficit; energy balance; energy availability; physical activity
MeSH Terms: conditions — Relative Energy Deficiency in Sport; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy deficit (Experimental): Diet-induced 50% energy deficit (based on estimated average total daily energy expenditure) by allocation of pre-made meals and snacks over 7-days
  Interventions: Dietary Supplement: Controlled energy-deficit diet
- Energy surplus (Experimental): Diet-induced energy surplus (approximately 500-1000kcal/day) achieved by allocation of additional snacks to be consumed on top of habitual free-living diet, to avoid inadvertent energy deficit
  Interventions: Dietary Supplement: Habitual diet with surplus snacks

INTERVENTIONS:
Dietary Supplement: Controlled energy-deficit diet — Participants receive a prepared diet providing approximately 50% of their estimated daily energy expenditure to induce a sustained energy deficit
  Other Names: Energy deficit
  Arms: Energy deficit
Dietary Supplement: Habitual diet with surplus snacks — Participants continue their normal diet with the addition of high-calorie snack items to achieve an approximate daily energy surplus
  Other Names: Energy surplus
  Arms: Energy surplus

SUMMARY:
Recent research has suggested that increasing levels of physical activity are associated with a reduction in the independent components that contribute to total energy expenditure (such as resting metabolic rate and non-exercise movement) - this occurs to conserve energy required for physical activity where energy provision becomes scarce. There are potential deleterious health and performance consequences of a reduced energy supply to fundamental metabolic processes, putting individuals regularly undertaking high levels of physical activity, such as endurance athletes, at risk. However, this association is largely based on observational data in only moderately active populations, and it is currently unclear what role energy balance status and biological sex has on this relationship.

This research intends to address these unknowns by assessing the impact of diet-induced manipulation of energy balance (conditions of energy deficit and energy surplus) in individuals undertaking habitually high levels of physical activity on independent components of total energy expenditure (resting metabolism, exercise and non-exercise movement).

Male and female athletes conducting regular moderate-to-high training volumes will undertake a randomised crossover study with a 7-day state of energy deficit and a 7-day state of energy surplus. Participants will continue to live and train as normal, but their diet will be controlled by specific food provision over the intervention periods in order to facilitate both conditions. Independent components of energy expenditure, markers of health, metabolism and performance will be measured to allow for comparison of conditions.

DETAILED DESCRIPTION:
People with very active lifestyles such as athletes, dancers, and military personnel, need to eat a lot of food to make up for the large amount of energy they burn. If they don't match their food intake to their energy needs, they may enter a state of 'energy deficit'. This means their bodies are burning more calories than they're taking in, which can lower performance, increase the risk of injuries and illnesses, and potentially harm overall health.

Traditional scientific understanding assumes that more doing physically activity leads to burning more calories (the 'additive' model). However, newer studies suggest that the body might have built-in safeguards to limit how many total calories it burns, no matter how much a person exercises. This idea (the 'constrained' model) proposes that when people exercise more, their bodies might compensate by slowing down other metabolic processes to keep overall energy use within a certain range. Although this mechanism could help the body conserve energy, it may also mean that essential functions (like immune system support and reproductive function) can become impaired.

Most research on energy deficit so far has focused on people with normal or moderate levels of physical activity. Because extremely active people experience far higher daily energy demands, the 'constrained' mechanisms could manifest differently or to a greater degree and the negative health and performance consequences might be more severe. There is also limited knowledge about how quickly these changes in energy use begin and how they affect important processes at the cellular level, such as muscle mitochondrial function or immune cell health.

This study aims to fill these gaps by measuring total energy use (and its separate parts) in highly active individuals under two conditions: when participants eat enough to cover their energy demands and when participants are purposely in an energy deficit (intentionally eating less than they need). One of our main goals is to measure changes in resting metabolic rate (RMR), which is the energy the body uses at rest to keep vital functions going. Investigators will also examine cellular changes by looking at indicators like immune cell function to see how these might help us detect early signs of harmful energy shortages.

By understanding whether, and to what extent, the body's energy use is 'constrained', investigators can develop better guidelines to help very active individuals avoid unhealthy energy deficits. Ultimately, this research could improve both performance and long-term health for athletes, military personnel, dancers, and anyone else who regularly exercises at high levels.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified endurance-trained sport participants
* Training volume: >7 hours per week endurance training
* Training frequency: at least 5 days per week

Exclusion Criteria:

* Diagnosis of Relative Energy Deficiency in Sport (REDs)
* Active eating disorder (EDE-Q)
* Active flare of a chronic disease (e.g. inflammatory bowel disease)
* Type 1 or 2 diabetes mellitus
* Untreated or undergoing active treatment of anaemia (any cause)
* Current injury which precludes undertaking high volume endurance training
* Individuals following a habitual low-carbohydrate, high-fat diet
* Any medical diagnosis which precludes intense exercise (e.g. untreated cardiac arrhythmia)
* Allergy or intolerance to study foods
* Blood donation within preceding 8 weeks of study start date
* Use of medications that affect substrate utilisation (e.g. statins, corticosteroids, thyroxine, HRT)
* For females: current pregnancy, breastfeeding within past 6 months or post-menopausal
* Unable to undertake a treadmill running test
* Participation in any research study in the past 8 weeks
* Participation in a research study within the past year involving more than one DEXA scan
* Unable to provide informed consent due to impaired cognitive capacity or decision-making ability

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Resting metabolic rate (RMR) in kcal/day | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks.
  The effect of a 7-day period of energy expenditure-matched diet-induced energy deficit versus energy surplus on RMR. Measured via indirect calorimetry using the Douglas bag method. Expired gas will be collected in a seated, fasted state under thermoneutral conditions, and oxygen consumption and carbon dioxide production will be used to calculate energy expenditure.

SECONDARY OUTCOMES:
Total energy expenditure (from doubly labelled water) in kcal/day | Measured during both 7-day interventions starting at approximately week 4 and week 9.
Total energy expenditure ( from sum of independent components of energy expenditure) in kcal/day | Measured during both 7-day interventions starting at approximately week 4 and week 9
Peripheral blood mononuclear cell (PBMC) mitochondrial respiration | Measured pre- and post-exercise at visits 2/3 (pre- and post-intervention 1) and visits 4/5 (pre- and post-intervention 2), approximately weeks 4-12.
  Assessment of mitochondrial respiratory function in isolated PBMCs using high-resolution respirometry (Oroboros). Measures include basal (routine), leak, oxidative phosphorylation (OXPHOS), and electron transfer system (ETS) capacity states. Data will be used to assess changes in mitochondrial function in response to exercise and nutritional intervention. Units: pmol O₂·s-¹·10⁶ cells-¹ (picomoles of oxygen consumed per second per million PBMCs).
Sub-maximal exercise performance (during steady-state treadmill exercise) | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks.
  Running economy (oxygen consumption at a fixed submaximal speed, expressed as ml O₂·kg-¹·min-¹)
Free T3 in pmol/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks.
Interstitial glucose concentration in mmol/l | Measured during both 7-day interventions starting at approximately week 4 and week 9.
  Continuous glucose monitoring using Dexcom G7 reporting mean daily and daily variability in interstitial glucose concentration.
Bone mineral density (DEXA) | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks.
  Bone mineral density will be assessed using dual-energy X-ray absorptiometry (DEXA). DEXA will provide areal BMD (g/cm²).
Bone mineral density (pQCT) | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks.
  Bone mineral density will be assessed using peripheral quantitative computed tomography (pQCT) at the tibia. Measures will include volumetric BMD (vBMD) in mg/cm³ in cortical and trabecular compartments.
Subjective measures of fatigue | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks.
  Daily subjective fatigue will be assessed using the Hooper Index (fatigue subscale, 5-item 1-5 Likert scale). Higher scores indicate greater perceived fatigue.
  Units: Hooper Index: total score (5-25)
Sleep duration in h/night | Measured during both 7-day interventions starting at approximately week 4 and week 9.
  Accelerometer-dervied using arm-worn Actigraph LEAP device.
Non-exercise activity thermogenesis (NEAT) (estimated from ActiGraph LEAP device) in kcal/day | Measured during both 7-day interventions starting at approximately week 4 and week 9
Exercise energy expenditure (estimated from ActiGraph LEAP device) in kcal/day | Measured during both 7-day interventions starting at approximately week 4 and week 9
Sub-maximal exercise performance (during steady-state treadmill exercise) | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks
  Substrate utilisation (absolute in g·min-¹)
Sub-maximal exercise performance (during steady-state treadmill exercise) | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks
  Substrate utilisation (relative as % total energy expenditure)
Bone mineral density (pQCT) | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks
  Cross-sectional area in mm²
Bone mineral density (pQCT) | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks
  Strength-strain index in mm³
Subjective measures of fatigue | Measured at lab visits 1-5 (baseline and pre- and post-interventions) from 0 to 12 weeks.
  Daily subjective fatigue will be assessed using the Fatigue Assessment Scale (FAS), a 10-item validated questionnaire scored from 10 to 50. Higher scores indicate greater perceived fatigue.
  Units: total score (10-50).
Total testosterone in nmol/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
Free testosterone in pg/mL | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
cortisol in nmol/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
IGF-1 in ng/mL | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
leptin in ng/mL | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
Female-specific hormones: oestradiol in pmol/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
Female-specific hormones: FSH in IU/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
Female-specific hormones: LH in IU/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
Inflammatory markers: interleukin-6 (IL-6) in pg/mL | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
high-sensitivity C-reactive protein (hsCRP) in mg/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
ferritin in µg/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
serum iron in µmol/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
transferrin in g/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
total iron binding capacity (TIBC) in µmol/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
transferrin saturation as a percentage | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
soluble transferrin receptor in mg/L | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
hepcidin in ng/mL | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
Lipid markers: total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides in mmol/L; non-esterified fatty acids (NEFA) in mmol/L; and glycerol in µmol/L. | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks
HbA1c will be reported in both % (DCCT-aligned) and mmol/mol (IFCC standard). | Measured at lab visits 2-5 (pre- and post-interventions) from 4 to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided